CLINICAL TRIAL: NCT01500980
Title: Infection-Treatment-Vaccination for Plasmodium Falciparum
Brief Title: Malaria Challenge in Healthy Volunteers
Acronym: ITV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MC-003
Record Dates: First submitted 2011-12-19; First posted 2011-12-29 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Malaria
Keywords: malaria; challenge; P. falciparum; prevention
MeSH Terms: conditions — Malaria | interventions — Chloroquine; Primaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Pilot Phase (Experimental): Pilot phase will include 6 subjects and will investigate the timing of PQ dosing relative to parasite exposure.
  Interventions: Biological: P. falciparum infection; Drug: Chloroquine; Drug: Primaquine
- Chloroquine, ITV, primaquine, malaria challenge (Experimental)
  Interventions: Biological: P. falciparum infection; Drug: Chloroquine; Drug: Primaquine
- Sporozoite negative vaccine (Active Comparator)
  Interventions: Drug: Chloroquine; Drug: Primaquine
- Primaquine placebo (Active Comparator)
  Interventions: Biological: P. falciparum infection; Drug: Chloroquine
- malaria challenge (No Intervention)

INTERVENTIONS:
Biological: P. falciparum infection — P. falciparum (NF54 strain) infection delivered by the bites of 12 - 15 infected A. stephensi mosquitos
  Arms: Chloroquine, ITV, primaquine, malaria challenge; Pilot Phase; Primaquine placebo
Drug: Chloroquine — Weekly chloroquine dosing (600 mg loading dose, 300 mg thereafter)
  Arms: Chloroquine, ITV, primaquine, malaria challenge; Pilot Phase; Primaquine placebo; Sporozoite negative vaccine
Drug: Primaquine — Primaquine (45 mg) on day 2 or 3 post ITV infection
  Arms: Pilot Phase
Drug: Primaquine — Primaquine (45 mg) on day 2 or 3 (pending results of pilot study) post ITV infection
  Arms: Chloroquine, ITV, primaquine, malaria challenge; Sporozoite negative vaccine

SUMMARY:
The purpose of this study is to determine if sterile, protective immunity to malaria can be induced by malaria parasite exposure limited to the early liver stage of the parasite lifecycle.

DETAILED DESCRIPTION:
This randomized, partial double-blind, placebo-controlled phase 1 study is designed to evaluate whether sterile protective immunity to P. falciparum can be induced by wild-type (non-attenuated) sporozoite immunizations when exposure is limited to sporozoite and early liver stage of the parasite life cycle and at a low dose sporozoite inoculum relative to other whole parasite vaccination models using live attenuated P. falciparum parasites (e.g. irradiated sporozoites). A secondary objective of the study is to evaluate newly identified antigens as potential targets of an immune response preferentially induced in individuals protected by whole sporozoite vaccination. Once identified as immune targets, these antigens can then be prioritized for subunit vaccine development. Subjects will be closely monitored for signs and symptoms of malaria and/or drug toxicity throughout the study.

A total of 36 healthy, malaria-naive adult subjects will be enrolled in the study. Six subjects will be randomized to the Pilot Phase (Arm 1), 24 to the Main ITV Phase (Arms 2, 3, and 4), and six subjects will be randomized for challenge control (Arm 5) to start on the day of challenge of the Challenge Phase.

Subjects in Arms 1-4 will receive three episodes of ITV immunization and a subsequent challenge with homologous P. falciparum sporozoites in the absence of chemoprophylaxis. The ITV immunization in this study consists of:

1. Experimental infection with wild-type (non-attenuated) NF54 strain P. falciparum sporozoites delivered by the bites of 12 - 15 infected A. stephensi mosquitoes (ITV infection) administered in conjunction with
2. Causal prophylaxis with PQ or placebo, timed to eliminate parasites early in the liver stage of development, after hepatocyte invasion but prior to maturation and release into the bloodstream, and
3. Continuous suppressive prophylaxis with the blood-stage antimalarial drug CQ to prevent development of patent parasitemia and clinical malaria.

The study includes a Pilot Phase because the timing of PQ dosing relative to parasite exposure is critical to the efficacy of PQ as causal prophylaxis yet still allowing for maximized antigenic exposure to liver-stage parasites. The Pilot Phase will compare the prevention of blood-stage parasitemia by PQ administered two days vs. three days after a single ITV infection. Based on protection data from the Pilot Phase, a dosing algorithm will be used to determine timing of the PQ dose for the Main ITV Phase.

In the Challenge phase, which occurs after the three ITV events, sterile protective immunity will be assessed by challenge with homologous P. falciparum sporozoites in the absence of chemoprophylactic drugs. Five weeks after stopping chemoprophylaxis, subjects will undergo experimental P. falciparum infection by the bites of five infective mosquitoes and will be closely monitored for signs and symptoms of malaria in a hotel setting.

Subjects who develop patent parasitemia will be immediately treated with a standard dose of Malarone and withdrawn from the study. Treated subjects will continue to be monitored with daily blood smears until three consecutive daily blood smears are negative and any residual symptoms of malaria are mild or resolved.

Subjects are closely monitored throughout the study for solicited and unsolicited adverse events related to any part of the ITV immunization. The study is expected to last 4 to 9 months depending on which the subject is assigned, and may have up to 64 scheduled study visits during the time period.

Subjects will be followed in the clinic for 35 days after the challenge and a follow up phone call will be conducted at six months after the challenge. In an effort to evaluate the duration of an immune response to ITV, all subjects will be invited to return for optional evaluations at three and six months post challenge.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant females age 18 to 50 years
* Good general health status as demonstrated by medical history, physical exam, and screening laboratory test performed within 90 days of enrollment
* Ability and willingness to provide informed consent
* No laboratory evidence of hematologic, hepatic, or renal disease
* Assessment of Understanding questionnaire completed and passed prior to enrollment
* Reliable access to the clinical trials centers and availability to participate for duration of study
* If the subject is biologically female and of reproductive potential she must agree to consistent pregnancy prevention

Exclusion Criteria:

* Recent travel to a malaria endemic area within 6 months of enrollment
* Planned travel to a malaria endemic area during the study period
* History of confirmed malaria diagnosis on peripheral blood smear
* Anticipated use during the study period, or use within the following periods prior to enrollment:

  1. Investigational malaria vaccine at any time
  2. Malaria chemoprophylaxis within 6 months
  3. Chronic systemic immunosuppressive medications within 6 months
  4. Blood products or immunoglobulins within 120 days
  5. Investigational product or vaccine within 30 days
  6. Systemic antibiotics with antimalarial effects within 30 days
  7. Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to each ITV infection and challenge
  8. Medications known to interact with primaquine, chloroquine or atovaquone/proguanil (only during the study period)
* History of:

  1. Sickle cell disease, sickle cell trait, or other hemoglobinopathies
  2. Splenectomy or functional asplenia
  3. Systemic anaphylaxis
  4. Gelatin allergy
  5. Severe allergic reactions to mosquito bites of study drugs
  6. Documented history of chronic or active neurologic disease
  7. Psoriasis or porphyria
  8. Ocular diseases including retinopathy or visual field defects
* Glucose 6 phosphate dehydrogenase (G6PD) deficiency
* Clinically significant medical condition, physical examination findings, other clinically significant abnormal laboratory results, or past medical history that may have clinically significant implications for current health status in the opinion of the Investigator.
* Weight <55 kg or >90 kg; body mass index (BMI) <18.5% or >31%
* History of known active cardiac disease or stroke
* Clinically significant abnormal screening electrocardiogram (ECG)
* Moderate or high risk for coronary heart disease (CHD) based on NHANES I cardiovascular risk assessment
* Acute illness at the time of enrollment
* Pregnant or nursing female
* Infection with HIV, Hepatitis B, Hepatitis C
* Psychiatric condition that precludes compliance with the protocol
* Suspected or known current alcohol or drug abuse
* Any other finding that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a subject's ability to give informed consent, or increase the risk of having an adverse outcome from participating in the study
* Clinical trial staff with direct involvement in the conduct of the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Microscopic evaluation of peripheral blood smears | Up to 182 days
  Detection for evidence of patent parasitemia and time to parasitemia following challenge with homologous P. falciparum sporozoites in subjects with confirmed exposure to P. falciparum sporozoites and early liver stage parasites only
qRT-PCR | Up to 182 days
  qRT-PCR evaluation for detection of subpatent parasitemia following a single episode of ITV
Number of subjects with adverse events | up to 182 days
  Occurrence of solicited and unsolicited adverse events (AEs) and serious adverse events (SAEs) during the study period

SECONDARY OUTCOMES:
ELISA | up to 182 days
  Humoral immune responses pre-/post- ITV and subsequent challenge by binding ELISA for antibodies to P. falciparum liver stage, blood stage, and pre-erythrocytic antigens.
IFN-y ELISPOT | up to 182 days
  Evaluation of cell-mediated immune responses to P. falciparum liver-stage and pre-erythrocytic antigens pre-/post- ITV and subsequent challenge by (IFN-y) ELISPOT assay on peripheral blood mononuclear cells
ICS assay | up to 182 days
  Detection of cell-mediated immune responses pre-/post- ITV and subsequent challenge by ICS assay for P. falciparum pre-erythrocytic antigens on peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Sara Healy, M.D. MPH, Principal Investigator — Seattle Biomedical Research Institution
Locations (1):
- Seattle Biomedical Research Institute's Malaria Clinical Trials Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Healy SA, Murphy SC, Hume JCC, Shelton L, Kuntz S, Van Voorhis WC, Moodie Z, Metch B, Wang R, Silver-Brace T, Fishbaugher M, Kennedy M, Finney OC, Chaturvedi R, Marcsisin SR, Hobbs CV, Warner-Lubin M, Talley AK, Wong-Madden S, Stuart K, Wald A, Kappe SH, Kublin JG, Duffy PE. Chemoprophylaxis Vaccination: Phase I Study to Explore Stage-specific Immunity to Plasmodium falciparum in US Adults. Clin Infect Dis. 2020 Sep 12;71(6):1481-1490. doi: 10.1093/cid/ciz1010. PMID 31621832